CLINICAL TRIAL: NCT03940482
Title: Time Restricted Eating As Treatment (TREAT) for Diabetes Mellitus: A Pre-Post 12 Week Study on the Effectiveness of Intermittent Fasting in Asians With Type 2 Diabetes Mellitus
Acronym: TREAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TREAT-DM-01
Record Dates: First submitted 2019-04-16; First posted 2019-05-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: TYPE 2 Diabetes Mellitus; Intermittent Fasting; Time Restricted Eating as Treatment (TREAT)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Intermittent Fasting | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Subjects will act as their own controls
  Interventions: Behavioral: Time Restricted Eating As Treatment (TREAT) for Diabetes.

INTERVENTIONS:
Behavioral: Time Restricted Eating As Treatment (TREAT) for Diabetes. — Participants will skip a meal every day and maintain a water only fast for 16 hours. A fasting diary is kept to track hours of fasting. Participants will follow this new pattern of eating for 12 weeks. They will visit the doctor's office at least 3 times in the course of the study and will be followed up with anthropometry (weight, BMI and waist circumference) and biochemical markers pertaining to Diabetes during the study visits. At 24 weeks, a follow up phone call will be made to check self-reported compliance to intermittent fasting.

SUMMARY:
Type 2 Diabetes Mellitus (DM) is a silent epidemic that affects 11.3% of Singaporeans. It has numerous clinical sequelae including macrovascular and microvascular disease. Nutritional therapy has been widely accepted as being safe and affordable as compared to pharmacotherapy. It is estimated that current nutritional therapy is able to reduce HbA1c levels by 1 to 2 percent under ideal circumstances. A weight loss of >5% is needed to have any significant beneficial effects on the levels of HbA1c, lipids, and blood pressure. This requires extensive modification of lifestyle, calorie restriction, regular exercise, and close supervision by health care professionals; impracticable for most patients. Intermittent Fasting that has been shown to be effective in improving the metabolic state of human subjects. The investigators ask if a simpler dietary regime based on time restricted eating would produce the necessary weight loss and good metabolic outcome.

In this pilot single arm pre-post study, 50 adult diabetic patients will be educated on Time Restricted Eating As Treatment (TREAT). Under this intervention, subjects will skip one meal a day and aim for a fasting period 16 hours a day. In the 8 hours where eating is permitted, subjects are encouraged to eat normally based on what is recommended for diabetic patients in usual care. Relevant clinical parameters, such as blood glucose control, lipid and triglyceride levels and anthropometry will be monitored over a 12-week period.

This study would have major clinical impact if it is found that TREAT can result in the improvement of cardiometabolic parameters and is practicable and sustainable in a real world setting.

DETAILED DESCRIPTION:
Nutritional therapy for diabetes mellitus is widely accepted as safe and affordable when compared to pharmacotherapy. However, the efficacy of the present state of nutritional therapy based on current recommendations is poor. It is estimated that nutritional therapy is able to reduce HbA1c levels by 1 to 2 percent under ideal circumstances. A weight loss of >5% is needed to have any significant beneficial effects on the levels of HbA1c, lipids, and blood pressure. This would require extensive modification of lifestyle, including calorie restriction, regular exercise, and close supervision by health care professionals. For the majority of patients, adherence to such a regime on a long-term basis is not achievable or practical.Considerable effort is required to educate and reinforce the complex behavioural changes needed. A simpler dietary regime that would produce the necessary weight loss and good metabolic outcome is needed.

Rationale for use of Intermittent Fasting as Nutritional Therapy: Practicability, Efficacy and Safety.

Intermittent fasting (IF) has been practiced by humans since ancient times, out of necessity and for religious purposes. Numerous regimens of intermittent fasting exist:

1. Alternate-day fasting, with either a total fast or restriction of energy 60-70% below estimated requirements on alternate days.
2. Modified Fasting Regimens (such as the 5:2 diet which involves severe energy restriction for 2 non-consecutive days in a week and ad libitum eating for the other 5 days), a variant of alternate-day fasting.
3. Time-restricted Feeding where intake is restricted to a pre-defined time window daily, and fasting occurs for 12-21 hours of the day.

There is experimental and evolutionary evidence across microbes and animals that such fasting improves cardiometabolic health and survival. In mice, the preservation of beta cell function occurs through the mechanism of autophagy during fasting, and survival is prolonged in bacteria, yeasts, worms and mice when fasting that has been attributed to an alternative ketone-body like energy source during periods of caloric deprivation. The mechanisms of action proposed are that fasting triggers adaptive cellular stress responses, resulting in an enhanced ability to cope with more severe stress and counteract disease processes. In addition, by protecting cells from DNA damage, suppressing cell growth and enhancing apoptosis of damaged cells, fasting could retard and/or prevent the formation and growth of cancers.

In humans, there is increasing evidence that intermittent fasting produces improvements in various metabolic parameters that are potentially beneficial to Type 2 Diabetics, such as improvements in glycaemic control, lipid profiles and weight loss. For example, Carter reported equivalent reductions in HbA1c in individuals with Type 2 diabetes with 12 weeks of Intermittent Energy Restriction (IER) or Continuous Energy Restriction (CER) which had been achieved with greater reductions in insulin medications within the IER group. Arnason demonstrated improved glycaemic control and weight in 10 community-dwelling middle-aged Type 2 Diabetic adults over a six week period in which subjects underwent Time-restricted feeding intervention for 2 weeks.

Other than glycaemic control, intermittent fasting also benefits other cardiometabolic parameters. Body fat, LDL-Cholesterol, Triglycerides and weight circumference were reduced with improvements in glucose metabolism in obese subjects in response to an alternate day modified fast. Glucose metabolism, reflected by decrease in fasting insulin, improved in non-obese subjects when subjected to 3 weeks of alternate day fasting.

Alternate day fasting has been associated with hunger, distraction with lower perceived work performance and lower mood reported across some of its' human studies.Modified Fasting Regimens, though they largely result in clinically and statistically significant weight loss of between 3.2-8.0% have up to 15% of participants reporting negative side effects, such as feeling cold, irritable, low energy levels or hunger.

Time-restricted Feeding (TRF), typically have daily fasting intervals of 12-21 hours per day. There were no mean changes in tension, depression, anger, vigor, fatigue or confusion when subjects of a crossover trial were consuming one meal a day as opposed to an isocaloric diet consumed as three meals a day. There is observational evidence from Ramadan studies of Diabetic patients that glycaemic control and lipid parameters improve over a 4-week fasting period. Only one cross-over controlled study in healthy middle-aged adults has reported on metabolic outcomes with Time-restricted Feeding. Stote et al. found both pro-atherogenic changes (increased LDL cholesterol) and anti- atherogenic changes (increased HDL cholesterol and decreased TG) following 8 weeks of limiting food intake to one evening meal. This might have been confounded by circadian variations of baseline and post-intervention blood measurements, that were taken in the morning and evening respectively. Thus far, there are no publications on interventional studies on Time-restricted Feeding in diabetics to the investigators' knowledge. Time-restricted Feeding appears to be the most practical and easy to learn regime among all the intermittent fasting variations.

The investigators decided to adopt TRF and make it into a standardized regime that requires the subject to aim for a continuous fasting duration of 16 hours per day. The instruction can be taught to patients in a 30 minute session and opportunistic reinforcements. This mimics a real world counselling encounter between a primary care physician and patient with diabetes mellitus. The investigators call this regime Time Restricted Eating As Treatment (TREAT). This 12-week study of TREAT in adult patients with Type 2 Diabetes Mellitus aims to explore if this simplified form of intermittent fasting can result in clinically and statistically significant reductions in weight, improved glycaemic control and metabolic parameters including hyperinsulinemia, with particular emphasis on an Asian population. Accordingly, the investigators plan to recruit 50 community dwelling type 2 diabetic patients and instruct them on TREAT in a clinic setting. Patients will then be followed up with anthropometry and biochemical markers pertaining to diabetes during the study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects (male or female) ≥ 21 to 80 years of age at Visit 1.
2. Subjects newly diagnosed with Type II diabetes mellitus (DM) who are solely on dietary control.
3. Ability to sign written informed consent before any study-specific procedure.
4. Subject is considered reliable and capable of adhering to protocol.
5. Subjects with Body Mass Index (BMI)≥ 23.5kg/m2.

Exclusion Criteria:

1. Subjects on Type II diabetes medication.
2. Subjects with any of the following medical conditions:

   * Congestive cardiac failure.
   * Stage 4 or worse chronic kidney disease (i.e. eGFR < 30 ml/min/1.73 m2)
   * Child's B or worse liver cirrhosis.
   * Any medical condition that in the opinion of the investigator could jeopardize or compromise the subject's ability to participate in the study.
3. Subject with previous or present history of eating disorder.
4. Subject not able to understand the informed consent form or fasting diary instructions.
5. Subject has participated in another study of an investigational medication or an investigational medical device within the last 30 days or is currently participating in these studies.
6. Subject is pregnant or lactating.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in glycaemic control of patients as measured by >= 5% reduction in glycosylated haemoglobin (HbA1C) over a 12 week period. | 12 weeks

SECONDARY OUTCOMES:
Change in glycaemic control of patients as measured by fasting glucose and 2 hour post prandial glucose over a 12 week period. | 12 weeks
  Fasting glucose would reduce significantly e.g. 0.5 mmol/L over a 12 week period. Post prandial glucose would decrease significantly e.g. 0.5 mmol/L over a 12 week period.
Change in Blood Pressure (BP) over a 12 week period. | 12 weeks
  Blood pressure would decrease significantly e.g. a systolic blood pressure drop of 7 mm Hg.
Change in Weight over a 12 week period. | 12 weeks
  Weight would reduce significantly e.g. 5% of initial body weight in kilograms.
Change in Body Mass Index (BMI) over a 12 week period. | 12 weeks
  Body Mass Index would decrease significantly e.g. 1 kg/m^2.
Change in Waist Circumference (WC) over a 12 week period. | 12 weeks
  Waist circumference would decrease significantly e.g. 3 centimeters.
Change in the lipid profiles of patients, namely Total Cholesterol (TC), High Density Lipoprotein (HDL), Low Density Lipoprotein (LDL), Triglycerides (TG), over a 12 week period. | 12 weeks
  Low density Lipoprotein would decrease significantly e.g. 0.5 mmol/L. Triglyceride experience a significant reduction e.g. 0.5 mmol/L.
Change in a levels of ketonemia (Serum Beta-Hydroxybutyrate 0.5-3.0 mmol/L) over a 12 week period. | 12 weeks
  Presence or absence of ketonemia evidenced by Serum Beta-Hydroxybutyrate 0.5-3.0 mmol/L over a 12 week period.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Kheng Hock, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital (Clinical Trials and Research Centre), Singapore, Singapore

REFERENCES:
- [Background] Franz MJ, Boucher JL, Evert AB. Evidence-based diabetes nutrition therapy recommendations are effective: the key is individualization. Diabetes Metab Syndr Obes. 2014 Feb 24;7:65-72. doi: 10.2147/DMSO.S45140. eCollection 2014. PMID 24591844
- [Background] Franz MJ, Boucher JL, Rutten-Ramos S, VanWormer JJ. Lifestyle weight-loss intervention outcomes in overweight and obese adults with type 2 diabetes: a systematic review and meta-analysis of randomized clinical trials. J Acad Nutr Diet. 2015 Sep;115(9):1447-63. doi: 10.1016/j.jand.2015.02.031. Epub 2015 Apr 29. PMID 25935570
- [Background] Patterson RE, Laughlin GA, LaCroix AZ, Hartman SJ, Natarajan L, Senger CM, Martinez ME, Villasenor A, Sears DD, Marinac CR, Gallo LC. Intermittent Fasting and Human Metabolic Health. J Acad Nutr Diet. 2015 Aug;115(8):1203-12. doi: 10.1016/j.jand.2015.02.018. Epub 2015 Apr 6. No abstract available. PMID 25857868
- [Background] Heilbronn LK, Smith SR, Martin CK, Anton SD, Ravussin E. Alternate-day fasting in nonobese subjects: effects on body weight, body composition, and energy metabolism. Am J Clin Nutr. 2005 Jan;81(1):69-73. doi: 10.1093/ajcn/81.1.69. PMID 15640462
- [Background] Halberg N, Henriksen M, Soderhamn N, Stallknecht B, Ploug T, Schjerling P, Dela F. Effect of intermittent fasting and refeeding on insulin action in healthy men. J Appl Physiol (1985). 2005 Dec;99(6):2128-36. doi: 10.1152/japplphysiol.00683.2005. Epub 2005 Jul 28. PMID 16051710
- [Background] Catenacci VA, Pan Z, Ostendorf D, Brannon S, Gozansky WS, Mattson MP, Martin B, MacLean PS, Melanson EL, Troy Donahoo W. A randomized pilot study comparing zero-calorie alternate-day fasting to daily caloric restriction in adults with obesity. Obesity (Silver Spring). 2016 Sep;24(9):1874-83. doi: 10.1002/oby.21581. PMID 27569118
- [Background] Williams KV, Mullen ML, Kelley DE, Wing RR. The effect of short periods of caloric restriction on weight loss and glycemic control in type 2 diabetes. Diabetes Care. 1998 Jan;21(1):2-8. doi: 10.2337/diacare.21.1.2. PMID 9538962
- [Background] Liu H, Javaheri A, Godar RJ, Murphy J, Ma X, Rohatgi N, Mahadevan J, Hyrc K, Saftig P, Marshall C, McDaniel ML, Remedi MS, Razani B, Urano F, Diwan A. Intermittent fasting preserves beta-cell mass in obesity-induced diabetes via the autophagy-lysosome pathway. Autophagy. 2017;13(11):1952-1968. doi: 10.1080/15548627.2017.1368596. Epub 2017 Nov 25. PMID 28853981
- [Background] Longo VD, Mattson MP. Fasting: molecular mechanisms and clinical applications. Cell Metab. 2014 Feb 4;19(2):181-92. doi: 10.1016/j.cmet.2013.12.008. Epub 2014 Jan 16. PMID 24440038
- [Background] Harvie M, Howell A. Potential Benefits and Harms of Intermittent Energy Restriction and Intermittent Fasting Amongst Obese, Overweight and Normal Weight Subjects-A Narrative Review of Human and Animal Evidence. Behav Sci (Basel). 2017 Jan 19;7(1):4. doi: 10.3390/bs7010004. PMID 28106818
- [Background] Carter S, Clifton PM, Keogh JB. The effects of intermittent compared to continuous energy restriction on glycaemic control in type 2 diabetes; a pragmatic pilot trial. Diabetes Res Clin Pract. 2016 Dec;122:106-112. doi: 10.1016/j.diabres.2016.10.010. Epub 2016 Oct 19. PMID 27833048
- [Background] Arnason TG, Bowen MW, Mansell KD. Effects of intermittent fasting on health markers in those with type 2 diabetes: A pilot study. World J Diabetes. 2017 Apr 15;8(4):154-164. doi: 10.4239/wjd.v8.i4.154. PMID 28465792
- [Background] Klempel MC, Kroeger CM, Varady KA. Alternate day fasting (ADF) with a high-fat diet produces similar weight loss and cardio-protection as ADF with a low-fat diet. Metabolism. 2013 Jan;62(1):137-43. doi: 10.1016/j.metabol.2012.07.002. Epub 2012 Aug 11. PMID 22889512
- [Background] Patterson RE, Sears DD. Metabolic Effects of Intermittent Fasting. Annu Rev Nutr. 2017 Aug 21;37:371-393. doi: 10.1146/annurev-nutr-071816-064634. Epub 2017 Jul 17. PMID 28715993
- [Background] Harvie M, Wright C, Pegington M, McMullan D, Mitchell E, Martin B, Cutler RG, Evans G, Whiteside S, Maudsley S, Camandola S, Wang R, Carlson OD, Egan JM, Mattson MP, Howell A. The effect of intermittent energy and carbohydrate restriction v. daily energy restriction on weight loss and metabolic disease risk markers in overweight women. Br J Nutr. 2013 Oct;110(8):1534-47. doi: 10.1017/S0007114513000792. Epub 2013 Apr 16. PMID 23591120
- [Background] Harvie MN, Pegington M, Mattson MP, Frystyk J, Dillon B, Evans G, Cuzick J, Jebb SA, Martin B, Cutler RG, Son TG, Maudsley S, Carlson OD, Egan JM, Flyvbjerg A, Howell A. The effects of intermittent or continuous energy restriction on weight loss and metabolic disease risk markers: a randomized trial in young overweight women. Int J Obes (Lond). 2011 May;35(5):714-27. doi: 10.1038/ijo.2010.171. Epub 2010 Oct 5. PMID 20921964
- [Background] Carlson O, Martin B, Stote KS, Golden E, Maudsley S, Najjar SS, Ferrucci L, Ingram DK, Longo DL, Rumpler WV, Baer DJ, Egan J, Mattson MP. Impact of reduced meal frequency without caloric restriction on glucose regulation in healthy, normal-weight middle-aged men and women. Metabolism. 2007 Dec;56(12):1729-34. doi: 10.1016/j.metabol.2007.07.018. PMID 17998028
- [Background] Al-Shafei AI. Ramadan fasting ameliorates oxidative stress and improves glycemic control and lipid profile in diabetic patients. Eur J Nutr. 2014 Oct;53(7):1475-81. doi: 10.1007/s00394-014-0650-y. Epub 2014 Jan 19. PMID 24442382
- [Background] Stote KS, Baer DJ, Spears K, Paul DR, Harris GK, Rumpler WV, Strycula P, Najjar SS, Ferrucci L, Ingram DK, Longo DL, Mattson MP. A controlled trial of reduced meal frequency without caloric restriction in healthy, normal-weight, middle-aged adults. Am J Clin Nutr. 2007 Apr;85(4):981-8. doi: 10.1093/ajcn/85.4.981. PMID 17413096